CLINICAL TRIAL: NCT06148467
Title: Incidence of Reverse Trigger Phenotypes and Response to Ventilatory Adjustments in Patients With ARDS
Brief Title: Reverse Trigger Phenotypification and Response to Ventilatory Adjustments
Acronym: RT-CHASERS
Status: Recruiting | Type: Observational
Sponsor: Hospital Civil de Guadalajara (Other)
Responsible Party: Principal Investigator, Miguel Á Ibarra-Estrada, MD, Hospital Civil de Guadalajara
Other Study IDs: 260/22
Record Dates: First submitted 2023-11-19; First posted 2023-11-28 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Reverse Trigger; Acute Respiratory Distress Syndrome; Mechanical Ventilation
Keywords: Reverse trigger; Acute Respiratory Distress Syndrome; Dyssynchony; Mechanical Ventilation
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this prospective observational study is to describe the incidence of reverse trigger (RT) in mechanically ventilated patients with diagnosis of acute respiratory distress syndrome (ARDS).

The main questions it aims to answer are:

* Real incidence of RT based on continuous monitoring
* The response to mechanical ventilatiory adjustments Participants will be included as soon as neuromuscular blockers (NMB)/sedation is stopped or in case of spontaneous respiratory efforts detection, whatever happens first. Continuous monitoring will be performed by esophageal manometry until switch to a pressure support (spontaneous) mode, restart of deep sedation/neuromuscular blockers by medical indication, or death.

In order to allow detection of possible RT in patients with ongoing sedation/NMB, mechanical ventilator waveforms will be screened every 1-2 hours by investigators and critical care physicians with at least 1 year of specific training in detection of dyssynchronies.

DETAILED DESCRIPTION:
Measurements:

An esophageal catheter for manometry will be placed as usual practice with confirmation of adequate position with the Baydur's occlusion test before recordings. An independent flow sensor and pressure transducer will be placed and connected to a laptop computer to obtain real-time monitoring along with continuous recordings, which then will be off-line analyzed by two experts, for confirmation of RT and characterization.

Data collection:

Main cause of the acute respiratory failure and days on mechanical ventilation until enrollment will be collected as well as demographic characteristics, including APACHE II, SOFA and the previous requirement of prone positioning therapy.

At identification of the RT, drugs for sedation and analgesia, time from initiation of mechanical ventilation to RT identification and blood gas analysis will be recorded. Ventilatory settings will also be collected, including the control variable of the ventilatory mode (volume or pressure), respiratory rate, received tidal volume in ml/kg of predicted body weight, maximum inspiratory flow, ratio of partial arterial oxygen pressure (pO2) to fraction of inspired oxygen (FiO2), driving pressure and (positive end-expiratory pressure (PEEP). Data about esophageal pressure related to RT will also be recorded, including the magnitude of pressure swing, phase angle, coefficient of variation, RT phenotype, entrainment ratio and the presence of breath stacking.

Patient-centered outcomes including length of mechanical ventilation, intensive care and hospital length of stay, and mortality will be followed-up until 60 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ARDS according to the Berlin criteria and added New Global Definition 2023
* Mechanical ventilation

Exclusion Criteria:

* <18 years
* Tracheostomy status
* Pneumothorax
* Tube thoracostomy with air leaks

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated patients with acute respiratory distress syndrome.
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of reverse trigger | 60 days
  Proportion of patients who developed reverse trigger

SECONDARY OUTCOMES:
Days of mechanical ventilation | 60 days
  Days of mechanical ventilation
ICU length of stay | 60 days
  Days from ICU admission to discharge to wards
Mortality | 60 days
  Rate of deceased patients in percentage

OTHER OUTCOMES:
Duration of RT | 60 days
  Total time of presence of RT
Phenotypes of RT | 60 days
  Rate of the different phenotypes according to cycle initiation and termination of patient's respiratory effort
Intensity of breathing efforts | 60 days
  Intensity of respiratory efforts as measured by esophageal manometry
Association with severity | 60 days
  Association of RT with lung disease severity as measured by pO2:FiO2 ratio
Response to ventilatory adjustments | 60 days
  Change in RT characteristics after changing ventilatory settings

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Ibarra Estrada, MD, Principal Investigator — Hospital Civil Fray Antonio Alcalde
Locations (1):
- Hospital Civil Fray Antonio Alcalde, Guadalajara, Mexico

IPD SHARING:
Plan to Share IPD: Undecided